CLINICAL TRIAL: NCT06039839
Title: Use of a Double-layered Collagen Matrix for Preservation of the Maxillary Tuberosity Area Upon Free Connective Tissue Graft Harvesting
Brief Title: Using of Collagen Matrix for Maxillary Tuberosity Donor Area Preservation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI-03
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Soft Tissue Atrophy
Keywords: connective tissue graft; xenogeic collagen matrix; increasing of soft tissue thickness; dental implant; soft tissue augmentation; donor site

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first group (Active Comparator): Healing of the donor area will be accomplished without the use of collagen matrix
  Interventions: Procedure: Closure of the donor area after CTG harvesting without the use of collagen matrix
- second group (Experimental): Closure of the wound defect in the donor area in the region of the maxillary tuberosity will be carried out after CTG harvesting with the use of collagen matrix
  Interventions: Procedure: Closure of the donor area after CTG harvesting with collagen matrix

INTERVENTIONS:
Procedure: Closure of the donor area after CTG harvesting without the use of collagen matrix — 1. Incision the mucosa at the alveolar ridge, mucosal-periosteal flap elevation, placement of the dental implant
  2. Harvesting of free connective tissue graft from the maxilla tuberosity area and it's fixation to the vestibular mucosal-periosteal flap, tight suturing of the wound in the recipient area
  3. Suturing of the wound in the donor site.
  Arms: first group
Procedure: Closure of the donor area after CTG harvesting with collagen matrix — 1. Incision the mucosa at the alveolar ridge, mucosal-periosteal flap elevation, placement of the dental implant
  2. Harvesting of free connective tissue graft from the maxilla tuberosity area and it's fixation to the vestibular mucosal-periosteal flap, tight suturing of the wound in the recipient area
  3. Adaptation of sterile collagen matrix to the donor site
  4. Suturing of the wound in the donor site
  Arms: second group

SUMMARY:
An interventional prospective randomised clinical trial (RCT) in parallel groups is planned. The sample size was 30 patients who will be randomly divided into two groups based on the surgical procedure. The first group is the healing of the donor zone after SCTG harvesting without filling the wound with collagen matrix. The second group is the wound defect closure in the donor area using the collagen matrix "FibroMATRIX" (LLC "Cardioplant", Russia; registration in Russia 20/05/2019 No FSZ 2019/83671). Changes in volumetric parameters of the maxillary tuberosity area after CTG harvesting, severity of pain, postoperative edema, bleeding, analgesic intake and quality of life in the postoperative period will be assessed.

DETAILED DESCRIPTION:
The aim of this study is to perform a comparative analysis of the effectiveness of using a double-layer collagen matrix to preserve the parameters of the donor area in the region of the maxillary tuberosity versus healing of the wound surface without its use. Examination and treatment of patients will be carried out on the basis of the Department of Surgical Dentistry of the E.V. Borovsky Institute of Dentistry of I.M. Sechenov First Moscow State Medical University.

The object of the study will be patients with an inclusion defect on the maxilla or mandible within 1-2 teeth combined with a soft tissue thickness deficiency in the area of dental implants (< 2 mm) which requires mucosal augmentation operation. All patients will be randomly divided into two groups depending on the surgical procedure. In 1 group (n=15) the donor area will heal by secondary tension, and in 2 group (n=15) the collagen matrix "FibroMATRIX" will be used to close the wound defect in the donor area. The groups will be comparable in terms of gender and age characteristics. The randomisation of patients will be performed at the stage of surgical intervention as follows: after taking a free connective tissue graft and adapting the CTG to the recipient bed, an envelope with a randomly assigned method of donor area closure will be opened.

Patients in both groups will undergo dental implantation according to the standard protocol and healing abutment installation. In both groups of patients, a free connective tissue graft will be taken from the maxillary tuberosity and the autograft will be fixed to the vestibular full-thickness muco-periosteal flap with horizontal U-shaped sutures, followed by wound closure using simple interrupted sutures without tension.

Further, the collagen matrix "FibroMATRIX" (LLC "Cardioplant", Russia; registration in Russia 20/05/2019 No FSZ 2019/83671) will be adapted to the donor area for the patients of the 2 group, the patients of both groups will have to perform suturing of the wound surface using simple interrupted sutures.

In the postoperative period, standard antibacterial and anti-inflammatory therapy should be administered in combination with the use of topical antiseptics for daily care.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of written informed consent of the patient to participate in the study;
2. Age between 18 and 45 years;
3. Included defects on the maxilla or mandible within 1-2 teeth combined with soft tissue thickness deficiency in the area of dental implants (< 2 mm);
4. Teeth without periodontal pathology, probing depth should not exceed 3 mm across the entire dentoalveolar sulcus;
5. Satisfactory level of oral hygiene;
6. Absence of general diseases in the stage of exacerbation or decompensation

Non-inclusion criteria:

1. Patients who had previous harvesting of CTG from the same donor area;
2. Patients with impacted third molars in the donor area;
3. Presence of concomitant diseases in the stage of exacerbation or decompensation;
4. Patients with oncological diseases, as well as patients who have received radiotherapy and chemotherapy in the last 5 years;
5. Patients with a history of smoking for more than 10 years.

Exclusion Criteria:

1. Patient refusal of further participation in the study;
2. Pregnant and breastfeeding women;
3. Patients with blood coagulation disorders (haemophilia, Willebrand's disease, intake of anticoagulants);
4. Patients with diseases that impair soft tissue healing (insulin-dependent diabetes mellitus).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Changes in volumetric parameters of the maxillary tuberosity area after CTG harvesting | [Day 90 compared to the 0th day (initial value)]
  To carry out the measurement an optical impression will be taken using the Primescan intraoral scanner (Dentsply/SIRONA,Germany) before the operation and on the 90th day after the operation. Then, the stl files will be compared in the GOM Inspect software and the contour change will be evaluated at 3 equidistant points.

SECONDARY OUTCOMES:
Changes in volumetric parameters of the maxillary tuberosity area after CTG harvesting | [Day 180 compared to the 0th day (initial value)]
  To carry out the measurement an optical impression will be taken using the Primescan intraoral scanner (Dentsply/SIRONA,Germany) before the operation and on the 180th day after the operation. Then, the stl files will be compared in the GOM Inspect software and the contour change will be evaluated at 3 equidistant points.
Assessment of the severity of pain syndrome | [4 hours compared to the 0th day (initial value)]
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome was carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the severity of pain syndrome | [day 1 compared to the 0th day (initial value)]
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome was carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the severity of pain syndrome | [day 3 compared to the 0th day (initial value)]
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome was carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the severity of pain syndrome | [day 5 compared to the 0th day (initial value)]
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome was carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the severity of pain syndrome | [day 7 compared to the 0th day (initial value)]
  Visual Analogue Scale (VAS). Evaluation of the severity of pain syndrome was carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 3-4 - moderate pain; 5-6 - moderate-severe pain; 7-8 - severe pain; 9-10 - unbearable pain.
Assessment of the collateral edema | [day 1 compared to the 0th day (initial value)]
  Edema was clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues).
Assessment of the collateral edema | [day 3 compared to the 0th day (initial value)]
  Edema was clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues).
Assessment of the collateral edema | [day 5 compared to the 0th day (initial value)]
  Edema was clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues).
Assessment of the collateral edema | [day 7 compared to the 0th day (initial value)]
  Edema was clinically assessed by its volume (scores 0-2; 0 points - no edema, 1 point - moderate edema, 2 points - intense edema compared to the condition of adjacent tissues).
Assessment of bleeding | [day 1 compared to the 0th day (initial value)]
  Assessment of the presence of blood taste in the mouth using a scale where 0 - no taste, 1 - periodic taste, 2 - constant taste.
Assessment of bleeding | [day 3 compared to the 0th day (initial value)]
  Assessment of the presence of blood taste in the mouth using a scale where 0 - no taste, 1 - periodic taste, 2 - constant taste.
Assessment of bleeding | [day 5 compared to the 0th day (initial value)]
  Assessment of the presence of blood taste in the mouth using a scale where 0 - no taste, 1 - periodic taste, 2 - constant taste.
Assessment of bleeding | [day 7 compared to the 0th day (initial value)]
  Assessment of the presence of blood taste in the mouth using a scale where 0 - no taste, 1 - periodic taste, 2 - constant taste.
Assessment of consumption of analgesics | [day 1 compared to the 0th day (initial value)]
  Patients' analgesic consumption was assessed by estimating the number of packs of Nimesulide (100 mg) taken.
Assessment of consumption of analgesics | [day 3 compared to the 0th day (initial value)]
  Patients' analgesic consumption was assessed by estimating the number of packs of Nimesulide (100 mg) taken.
Assessment of consumption of analgesics | [day 5 compared to the 0th day (initial value)]
  Patients' analgesic consumption was assessed by estimating the number of packs of Nimesulide (100 mg) taken.
Assessment of consumption of analgesics | [day 7 compared to the 0th day (initial value)]
  Patients' analgesic consumption was assessed by estimating the number of packs of Nimesulide (100 mg) taken.
Assessment of the quality of life | [Day 0 (initial value)]
  The patient's quality of life was assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. The questionnaire consists of 14 questions that provide patient's self-reported measure of dysfunction, discomfort and disability arising from oral conditions. Each question is scored on a 5-point scale: 0 = never; 1 = hardly ever; 2 = occasionally; 3 = fairly often; 4 = very often/every day. The OHIP-14 total score can range from 0 to 56. Higher OHIP-14 scores indicate worse quality of life and lower scores indicate better quality of life.
Assessment of the quality of life | [Day 7 compared to the 0th day (initial value)]
  The patient's quality of life was assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. The questionnaire consists of 14 questions that provide patient's self-reported measure of dysfunction, discomfort and disability arising from oral conditions. Each question is scored on a 5-point scale: 0 = never; 1 = hardly ever; 2 = occasionally; 3 = fairly often; 4 = very often/every day. The OHIP-14 total score can range from 0 to 56. Higher OHIP-14 scores indicate worse quality of life and lower scores indicate better quality of life.
Assessment of the quality of life | [Day 90-93 compared to the 0th day (initial value)]
  The patient's quality of life was assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. The questionnaire consists of 14 questions that provide patient's self-reported measure of dysfunction, discomfort and disability arising from oral conditions. Each question is scored on a 5-point scale: 0 = never; 1 = hardly ever; 2 = occasionally; 3 = fairly often; 4 = very often/every day. The OHIP-14 total score can range from 0 to 56. Higher OHIP-14 scores indicate worse quality of life and lower scores indicate better quality of life.
Assessment of the quality of life | [Day 180-186 compared to the 0th day (initial value)]
  The patient's quality of life was assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. The questionnaire consists of 14 questions that provide patient's self-reported measure of dysfunction, discomfort and disability arising from oral conditions. Each question is scored on a 5-point scale: 0 = never; 1 = hardly ever; 2 = occasionally; 3 = fairly often; 4 = very often/every day. The OHIP-14 total score can range from 0 to 56. Higher OHIP-14 scores indicate worse quality of life and lower scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Ashurko, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
IPD Sharing is impossible because of the recommendation of the local ethics committee, the provision of data is possible upon receipt of an official request addressed to the chief researcher